CLINICAL TRIAL: NCT00902590
Title: A Genotype-Phenotype Urothelial Cancer Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Chicago (Other); Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-025
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Urothelial Cancer; Renal Pelvis Cancer; Ureter Cancer; Bladder Cancer
Keywords: renal pelvis; ureter; bladder; 09-025; Renal Pelvis, Ureter, Bladder Cancer
MeSH Terms: conditions — Ureteral Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cases will be invited to provide a saliva sample and tissue

GROUPS / COHORTS (2):
- 1: Patients with urothelial cancer
  Interventions: Other: saliva sample and questionaire
- 2: unrelated adults accompanying patients to clinic
  Interventions: Other: saliva sample, questionaire

INTERVENTIONS:
Other: saliva sample and questionaire — Urothelial Cancer Registry- Patients will complete a family history and urothelial cancer risk questionnaire, and will provide a buccal sample for germline DNA. If the cases have undergone germline sequencing as part of Protocol 12-245, they will not need to provide a buccal sample. If the cases have previously completed athe "the "Urothelial Baseline Questionnaire," in an MSKCC urology clinic they will not need to complete the urothelial cancer risk questionnaire.
  Groups: 1
Other: saliva sample, questionaire — Urothelial Cancer Registry- These participants will be requested to complete the risk factor questionnaire and to provide a saliva sample for DNA extraction.
  Groups: 2

SUMMARY:
This study is being done to create a registry to help us learn more about urinary and other cancers. This will let us look at large groups of people who do and do not have this kind of cancer.

The investigators will look at risk factors to learn more about how these impact cancer. The investigators will also look at genetic markers. These are genes that are found in a known place. They are often associated with a particular trait. If the gene changes in some way, it may predict cancer or response to treatment. The investigators will look for markers in your saliva.

This registry will help us develop better methods of:

Preventing these cancers. Diagnosing these cancers. Treating these cancers.

ELIGIBILITY:
Inclusion Criteria:

Urothelial Cancer Cases

* Must be ≥ 18 years of age AND
* Must have a diagnosis of urothelial cancer AND
* Must be an English-speaker

Non-Cancer Control Group

* Must be ≥ 18 years of age AND
* Must not have cancer or a personal history of cancer, with the exception of skin cancer. AND
* Must not be a blood relative of cases AND
* Must not be a blood relative of another control AND
* Must be an English-speaker

Family Member Control Group:

In select kindreds with a high prevalence of bladder cancer and/or very early onset bladder cancer, first- and second-degree family members of probands may be contacted by the MSKCC study team and invited to complete the questionnaire and submit a saliva sample.

* Must be ≥ 18 years of age AND
* Must be a blood relative of a case participant AND
* Must be an English-speaker

Exclusion Criteria:

* Have any condition, which in the opinion of the primary MSKCC clinician or investigators precludes their ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A member of the patient's treatment team, the protocol investigator, or a member of the research team at Memorial Sloan-Kettering Cancer Center (MSKCC) will identify potential research subjects. At MSKCC the following outpatient clinics will be used to recruit UC cases: Urology and Genitourinary Oncology. Patients and families may also be directly referred to the study team by any MSKCC physician, external physician, or by the family itself.
Sampling Method: Non-Probability Sample
Enrollment: 3519 (Actual)
Dates: Start 2009-05; Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Determine whether single nucleotide polymorphisms in regions discovered from whole genome scans, such as 8q24 & chromosome 3, & candidate genes, include NAT2 & GSTM1, prev found to be assoc with bladder ca risk, are assoc with UC in this study population | 2 years

SECONDARY OUTCOMES:
To determine whether single nucleotide polymorphisms in the genes and regions listed above are associated with outcomes after UC diagnosis in the population | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Iyer Gopakumar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org